CLINICAL TRIAL: NCT05328206
Title: Air Leak Test in Pediatric Intensive Care Unit : a Multicentric and Prospective Study
Brief Title: Air Leak Test In Pediatric Intensive Care Unit
Acronym: ALTIPICU
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Other Study IDs: APHP220207
Record Dates: First submitted 2022-03-04; First posted 2022-04-14 (Actual); Last update posted 2023-05-11 (Actual); Status verified 2023-05

CONDITIONS: Respiratory Distress; Upper Airway Obstruction
MeSH Terms: conditions — Dyspnea; Airway Obstruction | interventions — Standard of Care

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Standard of care for intubated children with a cuffed endotracheal tube (c-ETT)
  Interventions: Other: Standard of care for intubated children

INTERVENTIONS:
Other: Standard of care for intubated children — Patient ventilated through a cuffed endotracheal tube and having a cuff leak test prior extubation

SUMMARY:
Respiratory distress by upper airway obstruction (UAO) is the primary etiology of extubation failure in children hospitalized in pediatric intensive care unit (PICU).

This complication may require various invasive therapeutic which increase morbi-mortality and length of hospital stay.

Cuff leak test (CLT) measured prior extubation to predict post-extubation UAO has been widely used in adult. The test compared expired tidal volume with cuff inflated and cuff deflated in order to predict UAO.

Despite its frequent use in PICU, his predictive value to predict UAO in children is still poorly documented.

Therefore, we conducted the first multicentric, prospective study to evaluate the CLT as a predictor of post-extubation UAO in critically ill children.

The Primary objective is to assess the effectiveness of CLT in predicting severe respiratory distress by UAO within 48 hours of extubation in a critically ill children.

ELIGIBILITY:
Inclusion Criteria:

1. ≥ 2 day to < 18 years of age,
2. Ventilated through a cuffed endotracheal tube,
3. Expected duration of mechanical ventilation ≥ 24 hours,
4. Having a cuff leak test prior extubation,
5. Placed on the assist control setting during CLT,
6. No opposition from parents or patient

Exclusion Criteria:

1. Receiving mechanical ventilation via a tracheostomy,
2. Unplanned extubation,
3. Patient with long-term non-invasive ventilation (NIV),
4. History of upper airways pathology,
5. Surgery of upper airways less than 1 month old,
6. Limitations of medical care in place,
7. Parents or patient opposition,
8. Already been included in this study,
9. Not affiliated with social security.

Ages: 2 Days to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Child aged 2 days post-term to 18 years intubated with a cuffed endotracheal tube (c-ETT)
Sampling Method: Non-Probability Sample
Enrollment: 900 (Estimated)
Dates: Start 2022-10-05 (Actual); Primary Completion 2024-03-07 (Estimated); Study Completion 2024-04-03 (Estimated)

PRIMARY OUTCOMES:
Respiratory distress by post-extubation upper airway obstruction (UAO) | within 48 hours
  The respiratory distress will be assessed using the Westley score. The Westley score evaluates the severity of respiratory function by assessing five factors: level of consciousness, cyanosis, stridor, air entry, and retractions. A specific point values are given for each factor, and the final score sum has a range from 0 to 17. The greater the respiratory distress the more imminent the respiratory distress. Respiratory distress will be defined by a Westley score greater than or equal to 4 with a minimum of 1 for the "stridor" item, at the initiation of at least one of the following treatments (IVC, LNHD, NIV (CPAP, BiPAP or any other mode with two pressure levels), MV(reintubation or tracheotomy)).

SECONDARY OUTCOMES:
Cumulative incidence of return to mechanical ventilation (after re-intubation) | within 48 hours
Risk factors of severe respiratory distress (RD) | within 48 hours
  The respiratory distress will be assessed using the Westley score. The Westley score evaluates the severity of respiratory function by assessing five factors: level of consciousness, cyanosis, stridor, air entry, and retractions. A specific point values are given for each factor, and the final score sum has a range from 0 to 17. The greater the respiratory distress the more imminent the respiratory distress. Respiratory distress will be defined by a Westley score greater than or equal to 4 with a minimum of 1 for the "stridor" item, at the initiation of at least one of the following treatments (IVC, LNHD, NIV (CPAP, BiPAP or any other mode with two pressure levels), MV(reintubation or tracheotomy)).
Proportion of patients with intravenous corticosteroid therapy (IVC) | at inclusion
  Proportion of patients with intravenous corticosteroid therapy (IVC) in progress 12 hours prior to scheduled extubation, whether initiated for extubation or pre-extubation,
Predictive score for severe respiratory distress (RD) | within 48 hours
  The respiratory distress will be assessed using the Westley score. The Westley score evaluates the severity of respiratory function by assessing five factors: level of consciousness, cyanosis, stridor, air entry, and retractions. A specific point values are given for each factor, and the final score sum has a range from 0 to 17. The greater the respiratory distress the more imminent the respiratory distress. Respiratory distress will be defined by a Westley score greater than or equal to 4 with a minimum of 1 for the "stridor" item, at the initiation of at least one of the following treatments (IVC, LNHD, NIV (CPAP, BiPAP or any other mode with two pressure levels), MV(reintubation or tracheotomy)).
Median length of stay in paediatric intensive care | Up to 28 days

CONTACTS AND LOCATIONS:
Locations (19):
- France (19):
  - CHU Bordeaux Pellegrin, Bordeaux
  - Hôpital Haut-Lévêques, maladies cardio-vasculaires congénitales, Bordeaux
  - Hôpital Haut-Lévêques, réanimation chirurgicale cardiopédiatrique, Bordeaux
  - CHU Côte de Nacre, Caen
  - CHU Estaing, Clermont-Ferrand
  - Hôpital Raymond Poincaré, Garches
  - CHU Grenoble Alpes, Grenoble
  - CHU Bicêtre, Le Kremlin-Bicêtre
  - CHU Jeanne de Flandres, Lille
  - Hôpital Femme Mère Enfant HCL, Lyon
  - CHU de La Timone - AP-HM, Marseille
  - CHU Nancy, Nancy
  - CH Marie Lannelongue, Paris
  - Debré, AP-HP Nord, Paris
  - Necker, AP-HP Centre - Anesthésie, Paris
  - Necker, AP-HP Centre - Médecine intensive, Paris
  - Trousseau, AP-HP Est, Paris
  - CHU Toulouse, Toulouse
  - CHU Clocheville, Tours

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Lacarra B, Hayotte A, Naudin J, Maroni A, Geslain G, Poncelet G, Levy M, Resche-Rigon M, Dauger S. Air leak test in the Paediatric Intensive Care Unit (ALTIPICU): rationale and protocol for a prospective multicentre observational study. BMJ Open. 2024 Apr 30;14(4):e081314. doi: 10.1136/bmjopen-2023-081314. PMID 38688666